CLINICAL TRIAL: NCT01990703
Title: Randomized Controlled Trial of Early Versus Standard Postpartum Insertion of the Levonorgestrel IUD to Assess Breast Feeding Outcomes (BLIS - Breastfeeding Levonorgestrel IUD Study)
Brief Title: BLIS - Breastfeeding Levonorgestrel IUD Study
Acronym: BLIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Society of Family Planning (Other); University of New Mexico (Other)
Responsible Party: Principal Investigator, David Turok, M.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 62844
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Contraception
Keywords: Contraception; Birth Control; Levonorgestrel IUD; Mirena IUD
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early IUD Insertion Group (Experimental): Immediate post-placental placement of the levonorgestrel IUD
  Interventions: Drug: Levonorgestrel IUD
- Standard Postpartum Insertion Group (Active Comparator): Placement of the levonorgestrel IUD 4-6 weeks postpartum
  Interventions: Drug: Levonorgestrel IUD

INTERVENTIONS:
Drug: Levonorgestrel IUD — Timing of IUD insertion
  Other Names: Mirena

SUMMARY:
We are studying the effect of placing the levonorgestrel IUD (Mirena) immediately after birth on breastfeeding. Women who wish to have a levonorgestrel IUD placed after their birth, wish to breastfeed, and are willing to participate in the study will be randomly assigned to either get the IUD placed immediately after delivery of the baby and placenta or 4-6 weeks later. We do not believe there will be a difference in breastfeeding 8 weeks after delivery between those who get the IUD placed early or later.

DETAILED DESCRIPTION:
Increasing use of the levonorgestrel intrauterine device (LNG IUD) has become a cornerstone of U.S. efforts to decrease our nation's high rate of unplanned pregnancy. Many women initiate use of this method in the post partum period. The major advantage of immediate postplacental LNG IUD insertion is the prompt initiation of a highly effective contraceptive method at a time that does not interfere with the intense demands of newborn care, but any contraceptive method initiated in the postpartum period must not interfere with breastfeeding.

Our long-term goal is to understand the impact of hormonal contraceptives, initiated early in the postpartum period, on breastfeeding. The central hypothesis is that quality of breastfeeding is not negatively affected by progestin-only hormonal contraceptives.

We will pursue three specific aims comparing women randomized to immediate post-placental vs. delayed (4-6 week) postpartum LNG IUD insertion:

Aim #1: To determine breastfeeding continuation rates at 8 weeks in both groups Aim #2: To determine timing of lactogenesis in both groups Aim #3: To assess breastfeeding continuation, exclusivity, and satisfaction as well as continuation and satisfaction with the LNG IUD at 26 weeks postpartum in both groups

This proposal will support a non-inferiority RCT where participants will be randomly assigned to immediate postplacental insertion (within 10 minutes of placental delivery) or delayed postpartum insertion (4-6 weeks postpartum). This project will provide needed evidence on breastfeeding impact of early postpartum initiation of the LNG IUD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, 18-40 year old pregnant women
* Intend to breastfeed
* Desire the LNG IUD as their method of contraception
* Agree to be randomized to early versus standard postpartum insertion
* Have delivered a healthy term infant (37 weeks gestation)
* Willing to complete all study related procedures, visits and questionnaires

Exclusion Criteria:

* Chorioamnionitis
* Obstetric complications including transfusion
* Severe pregnancy induced hypertension
* Prolonged hospitalization
* Coagulopathy
* Liver disease
* Undiagnosed genital bleeding, or other relative contraindication to LNG IUD insertion (known or suspected pregnancy, uterine cavity abnormality, known, suspected, or history of breast cancer, or hypersensitivity to any of the components in the LNG IUD).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 285 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David K Turok, MD, Principal Investigator — University of Utah Department of Obstetrics & Gynecology
Locations (2):
- United States (2):
  - University of New Mexico, Albuquerque, New Mexico
  - University of Utah Health Sciences Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hopelian NG, Simmons RG, Sanders JN, Ward K, Jenkins SM, Espey E, Turok DK. Comparison of levonorgestrel level and creamatocrit in milk following immediate versus delayed postpartum placement of the levonorgestrel IUD. BMC Womens Health. 2021 Jan 21;21(1):33. doi: 10.1186/s12905-021-01179-7. PMID 33478494

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early IUD Insertion Group | Standard Postpartum Insertion Group
Started | 147 | 138
Completed | 108 | 93
Not Completed | 39 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early IUD Insertion Group | Standard Postpartum Insertion Group | Total
Number analyzed (Participants) | 147 | 138 | 285
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 147 | 138 | 285
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.6 (5.4) | 28.1 (5.6) | 28.4 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 138 | 285
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 147 | 138 | 285

OUTCOME MEASURES:

1. Primary Outcome: Breastfeeding Continuation Rates at 8 Weeks Postpartum
Description: To determine breastfeeding continuation rates at 8 weeks in women randomized to immediate post-placental vs. delayed (4-8 weeks) postpartum levonorgestrel IUD insertion.
Time Frame: 8 weeks postpartum
Population: 147 Early IUD Insertion participants at baseline drops to 112 at 8 weeks due to exclusions for medical complications (n=15), inability to provide immediate IUD (n=7) and loss to follow up (n=13). In the Standard Insertion group 138 at baseline drops to 102 at 8 weeks with medical comps (n=11), failure to receive IUD (n=24), and 1 loss to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Early IUD Insertion Group | Standard Postpartum Insertion Group
Number analyzed (Participants) | 112 | 102
Participants | 88 | 86

2. Secondary Outcome: Time to Lactogenesis Stage 2
Description: To evaluate potential delay in lactogenesis caused by immediate postpartum insertion of the LNG IUD.
Time Frame: First 5 days after birth
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Early IUD Insertion Group | Standard Postpartum Insertion Group
Number analyzed (Participants) | 125 | 103
Hours | 65.3 (25.7) | 63.6 (21.6)

ADVERSE EVENTS:
Arm/Group | Early IUD Insertion Group | Standard Postpartum Insertion Group
Serious Adverse Events (participants affected / at risk) | 1/147 | 0/138
Other Adverse Events (participants affected / at risk) | 1/147 | 0/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early IUD Insertion Group (N=147) | Standard Postpartum Insertion Group (N=138)
Suicidal behavior (Psychiatric disorders) | 1 (1) | 0 (0) — Participant hospitalized for suicidal behavior and lacerations after a history of severe recurrent depression.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early IUD Insertion Group (N=147) | Standard Postpartum Insertion Group (N=138)
Cholangitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant hospitalized for acute cholangitis with stone removal surgery performed.

LIMITATIONS AND CAVEATS:
Inability to blind, loss to follow-up, and lack of long-term infant and childhood outcomes. We had a smaller final sample than intended despite meeting enrollment goals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes